CLINICAL TRIAL: NCT06849999
Title: Evaluation of the Role of Kinesiophobia on Pain, Disability, and Quality of Life in Individuals with Chronic Neck Pain
Brief Title: Kinesiophobia in Chronic Neck Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSM PRH boyun
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Neck Pain; Kinesiophobia
Keywords: Chronic pain; Kinesiophobia; Disability; Quality of Life
MeSH Terms: conditions — Neck Pain; Kinesiophobia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, the effect of kinesiophobia on pain, disability, and quality of life in individuals with chronic neck pain will be evaluated. Neck pain is a common musculoskeletal disorder that can become chronic in some individuals. Kinesiophobia may lead to a reduction in physical activity due to fear of movement and re-injury, thereby increasing pain and disability. In this cross-sectional study, 57 participants will be assessed using the Visual Analog Scale (VAS), Tampa Scale for Kinesiophobia (TSK), Neck Disability Index (NDI), and the SF-36 Quality of Life Scale. Participants will be selected from individuals aged 18-59 who have experienced neck pain for at least 3 months, and those with a history of neurological disorders, spinal surgery, or pain treatment in the last 3 months will be excluded. This research aims to determine the effects of kinesiophobia on chronic neck pain, thereby contributing to the development of more effective treatment strategies. Written informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 59
* Patients of both genders experiencing neck pain for at least 3 months

Exclusion Criteria:

* Patients with neurological deficits
* Patients with any neurological disorder
* Patients with a history of spinal fractures, spinal tumors, or spinal infections
* Patients with a history of spinal surgery
* Patients with any congenital spinal anomaly
* Patients with vestibular disorders
* Patients taking antidepressant and antihypertensive medications
* Patients unwilling to participate in the study
* Patients who have received any pain treatment in the last 3 months
* Patients who have engaged in any strenuous physical activity within the 24 hours prior to the assessment

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Adults aged 18 to 59
  * Patients of both genders experiencing neck pain for at least 3 months
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
tampa kinesiophobia scale | 1 day
sf 36 | 1 day
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: pmr specialist, Principal Investigator — Liv hospital vadistanbul
Locations (1):
- Liv hospital Vadistanbul, Istanbul, Istanbul, Turkey (Türkiye)